CLINICAL TRIAL: NCT02550509
Title: Changes in Echogenicity and Muscle Stiffness in Elastography After Botulinum Toxin Injection a Spastic Muscle - A Monocentric Study
Brief Title: Changes in Echogenicity and Muscle Stiffness in Elastography After Botulinum Toxin Injection a Spastic Muscle
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties to include patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1301141
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: stroke; Botulinum toxin; Muscle alterations
MeSH Terms: conditions — Stroke | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with hemiplegia after stroke (Experimental): ultrasound echogenicity paraclinical assessment and elastography to patients with hemiplegia following stroke with an indication of injection of botulinum toxin into the triceps sural
  Interventions: Device: ultrasound echogenicity; Device: elastography

INTERVENTIONS:
Device: ultrasound echogenicity — ultrasound echogenicity to patient with stroke
Device: elastography — elastography to patient with stoke

SUMMARY:
Muscle alterations and modifications passive biomechanical properties that occur on a spastic muscle contribute to functional disorders involved in spasticity. Botulinum toxin (TB) A is the reference treatment of the focused spasticity, and muscle source structural and biomechanical changes, very little studied in humans, especially since it is not one possibility of easily and reliably paraclinical assessment injections consequences.

ELIGIBILITY:
Inclusion Criteria:

* A first stroke older than nine months (acute phase and subacute stroke).
* Hemiplegia cerebral vascular following this stroke.
* Hemiplegia with an overall motor deficit plegic lower limb muscle testing level less than or equal to 3 and associating a localized spasticity lower plegic member, on the plantar flexors, assessed by the upper Ashworth Scale or equal to 1 with an injection of botulinum toxin indication of the sural triceps.
* written consent.

Exclusion Criteria:

* Old stroke with motor impairment of the lower limb in the chronic stage.
* Concomitant muscle disease (eg myopathy, myositis ...).
* Patients who already received a botulinum toxin injection into the gastrocnemius muscles.
* Subjects with defibrillator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in muscular trophism | from baseline to 1 year
  Change in muscular trophism treated by botulinum toxin. Muscular trophism determined by a combined endpoint assessment of muscular echogenicity following scale Heckmatt I to IV, the measurement of the thickness in mm and angle pennation fascicular of medial and lateral gastrocnemius muscles to measured with an ultrasound scanner

CONTACTS AND LOCATIONS:
Overall Officials: PAul Calmels, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France